CLINICAL TRIAL: NCT04218682
Title: Narrating Their Story: Shadow's Edge Mobile Game Use to Enhance Resilience and Identity Formation Among Adolescent and Young Adult Survivors of Cancer
Brief Title: Shadows Edge Mobile Developing Resilience in Adolescent and Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Silicon Valley Community Foundation (Other)
Responsible Party: Principal Investigator, Bonnie Essner, PhD, Pediatric Psychologist, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB 2018-2137
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a waitlist randomized controlled study in which participants are randomly assigned to immediately begin to play the game (intervention) following enrollment versus wait 6 weeks to play the game following study enrollment. Participants will continue to receive all clinical care as usual throughout and following the study.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Game Use (Experimental): AYACS randomly assigned to this arm will immediately play the Shadow's Edge Game following enrollment for a duration of 7 weeks. Following the designated 7-week game-play period, they will continue to have access to the game. They will continue to receive all usual care health care throughout and following the study.
  Interventions: Behavioral: Shadow's Edge Mobile Application Gameplay
- Wait-List Comparison Group (No Intervention): AYACS randomly assigned to this arm will begin to play the Shadow's Edge game 7 weeks following enrollment. They will continue to receive all usual health care throughout and following the study.

INTERVENTIONS:
Behavioral: Shadow's Edge Mobile Application Gameplay — 6 weeks of individual, interactive game play of the Shadow's Edge mobile app.
  Arms: Immediate Game Use

SUMMARY:
This study evaluates the efficacy of an interactive mobile game, Shadow's Edge, on enhancing resilience, promoting identity development, and decreasing somatic symptoms among adolescent and young adult survivors of cancer.

DETAILED DESCRIPTION:
Approximately 80% of youth treated for cancer during childhood will survive long-term; however, the majority of adolescent and young adult cancer survivors (AYACS) report at least one chronic health condition. These medical and cognitive-psychological late effects can disrupt or interfere with continual adaptation to post-treatment life, thereby negatively impacting identity formation and inhibiting AYACS from seeking fulfilling academic, career, and social relationship experiences. The Shadow's Edge mobile app was created for adolescent and young adults with complex medical conditions as an enjoyable and engaging digital, first-person perspective game that uses principles of narrative and creative arts therapies to encourage youth to reflect on, and create brief, developmentally-relevant narratives about, their life experiences. In this trial, investigators will conduct a two-arm, waitlist randomized controlled trial to evaluate the effectiveness of the Shadow's Edge game in promoting resilience and identify formation among AYACS. Participants will be 175 AYACS who receive clinical care in a large, pediatric cancer survivorship program. Data will be collected from medical records, mobile game play statistics, participant narratives and art created in the game platform, and participant responses to standardized assessments. Information gathered through this study will be used to establish initial game efficacy and to lead to Shadow's Edge game enhancements that will further improve acceptability and effectiveness of the game. The ultimate goal of this project is to provide a freely accessible, enjoyable and engaging self-led game that may bolster resilience resources, improve quality of life, and promote identity formation among adolescents and young adults with complex medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent/young adults 13-24 years of age
* Adolescent/young adult English-speaking at a second grade level
* Parent/guardian English- or Spanish-speaking at a second grade level (for participants younger than 18 years of age)
* Patients with history of hematological malignancies (e.g., acute lymphoblastic leukemia) at maintenance phase of treatment or beyond or solid tumor patients (e.g., osteosarcoma) who have completed active treatment or cancer survivors with any form of malignancy history (excluding brain tumors) and are at least 2 years post-diagnosis of the malignancy
* Consistent access to a mobile phone and/or internet service

Exclusion Criteria:

* Brain tumor history
* History of moderate to severe neurodevelopmental disorder (e.g., autism spectrum disorder)

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Resilience | Baseline to 14-week follow-up
  Resilience will be measured by participant responses to the Brief Resilience Scale (BRS), a 6-item measure with response options on 5-point Likert scale ranging from "1, strongly disagree" to "5, strongly agree" and total scores ranging from 6 to 30 (higher scores indicating greater resilience).

SECONDARY OUTCOMES:
Perceived benefit and burden | Baseline to 14-week follow-up
  Perceived benefit and burden associated with the participant's cancer experience will be assessed with the 20-item Benefit and Burden Scale for Children. Participants rate statements on a five-point Likert scale, ranging from "1, not at all" to "5, very much, with higher scores on the 10-item Benefit scale indicating greater benefit-finding and higher scores on the 10-item Burden scale indicating greater perceived burden of the illness. Scores on each subscale range from 10 - 50.
Life meaning and purpose | Baseline to 14-week follow-up
  Meaning and purpose will be measured by the PROMIS Pediatric Meaning and Purpose Short Form-8. Items are rated on a five-point Likert scale ranging from "1, not at all" to "5, very much", with total scores ranging from eight to 40 (higher scores indicating greater sense of reason for living, goal direction, and hopefulness).
  ...scores range from 8 to 40 (higher scores indicate greater fear, anxious misery, and hyperarousal).
  The 8-item scale of depressive symptoms has scores ranging from 8 to 40 with higher scores indicating greater depressive symptoms. Total anxiety and total depression T-scores will be used in analyses.
Fatigue | Baseline to 14-week follow-up
  Fatigue over the past seven days will be measured with the PROMIS Pediatric Fatigue Short Form-10. Items are rated on a five-point Likert scale ranging from "1, never" to "5, almost always", with total scores ranging from 10 to 100 (higher scores indicating greater subjective feeling of tiredness, exhaustion and perception that fatigue interferes with daily function).
Pain Intensity | Baseline to 14-week follow-up
  Pain intensity over the past seven days will be measured with the PROMIS Pediatric Numeric Rating Scale - Pain Intensity, measured on an 11-point scale with anchors "0, No Pain" to "10, worst pain you can think of".
Positive affect | Baseline to 14-week follow-up
  Positive affect will be assessed by the PROMIS Pediatric Positive Affect Short Form-8. Items are rated on a five-point Likert scale ranging from "1, never" to "5, always", with total scores ranging from eight to 40 (higher scores indicating greater momentary positive affect, such as contentment, happiness, engagement, an excitement).
Depressive symptoms | Baseline to 14-week follow-up
  Depressive symptoms will be assessed by the PROMIS Pediatric Depressive Symptoms Short Form-8. Items are rated on a five-point Likert scale ranging from "1, never" to "5, almost always", with total scores ranging from eight to 40 (higher scores indicating greater negative mood, self-evaluation, and cognitions).
Anxiety | Baseline to 14-week follow-up
  Anxiety will be assessed by the PROMIS Pediatric Anxiety Short Form-8. Items are rated on a five-point Likert scale ranging from "1, never" to "5, almost always", with total scores ranging from eight to 40 (higher scores indicating greater fear, hyperarousal, and anxiety-associated somatic symptoms).
Self-identity after cancer | Baseline to 14-week follow-up
  Self-identity after cancer will be assessed with a four-item measure in which participants rate the degree to which they identify with four descriptions of relating to their past cancer experience. The five-point Likert scale ranges from "1, not at all" to "5, very much". Each item is used scored and used independently.
Identity status | Baseline to 14-week follow-up
  Identity status will be assessed via the 64-item Extended Objective Measure of Ego Identity Status-2. Participants rate each item on a 6-point Likert scale ranging from "1, strongly disagree" to "6, strongly agree", with total scores ranging from score of 64 to 384 (when measured on a continuous). Scores from this measure will be used to categorize participant identity status into one of four theoretically and empirically derived identity statuses and will also be used as a continuous variable, with higher scores indicating more mature identity status.
Daily pain intensity | Baseline to 14 week follow-up
  Daily pain intensity over the previous 24 hours will be measured with the PROMIS Pediatric Numeric Rating Scale - Pain Intensity v 1.0, measured on an 11-point scale with anchors "0, No Pain" to "10, worst pain you can think of". Daily pain intensity will be assessed over a 10-day period via daily diary.
Daily fatigue | Baseline to 14 week follow-up
  Daily fatigue over the past 24 hours will be measured with an 11-point 0 - 10 Numeric rating scale ranging from anchors of "not at all tired" to "very tired". Daily fatigue will be assessed over a 10-day period via daily diary.
Daily affect | Baseline to 14 week follow-up
  Daily affect over the past 24 hours will be assessed with Positive and Negative Affect Scale (PANAS), a 20-item measure in which participants rate the degree to which they have experienced each positive and negative emotion on a five-point Likert scale ranging from "1, Very slightly or Not at all" to "5, Extremely". Total scores for the Positive Affect Subscale and Negative Affect subscale range from 1 to 10. A "relative negative mood" index will be calculated for each participant whereby days in which the participant's negative affect score was greater than .5 standard deviations from that participant's 7-day mean negative affect scores will be designated as a "relative negative mood" day. Similarly, a "relative positive mood" index will be calculated for each participant whereby days in which the participant's positive affect score was greater than .5 standard deviations from that participant's 7-day mean positive affect scores will be designated as a "relative positive mood" day.
Sleep and sleep quality | Baseline to 14 week follow-up
  Each day for a consecutive 10-day period, participants will report the time they went to bed the previous night, the time they attempted to fall asleep, sleep onset delay, number of night awakenings, and that days' time that they awoke in the morning, time they got out of bed, the number of naps and duration of daytime sleep that day. They will also provide a subjective sleep quality rating using an 11-point 0 - 10 Numeric Rating Scale ranging from "0, extremely poor sleep" to "10, extremely good sleep".
Relative daily activity | Baseline to 14 week follow-up
  Each day for a consecutive 10-day period, participants' relative daily activity will be assessed with a form created for this study. Participants will rate the degree to which they engaged in five activities relative to their typical activity level. Responses are rated on an 11-point 0 - 10 NRS from "no, much less than usual" to "yes, much more time than usual".

OTHER OUTCOMES:
Intervention satisfaction | 14-weeks post-enrollment
  9-item measure created for this study, assessing participant enjoyment with the game intervention, elements of the game experience, and their perception that playing the game affected their emotions or behaviors. Range from 1=not at all to 5=very much

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Essner, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No